CLINICAL TRIAL: NCT01205360
Title: A Randomized, Control Study to Evaluate Dosing Strategies for Automated Mandatory Intermittent Boluses Technique for Epidural Labour Analgesia
Brief Title: Dosing Strategies for Automated Mandatory Intermittent Boluses Technique for Epidural Labour Analgesia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Pravara Institute of Medical Sciences University (Other)
Responsible Party: Dr.Mandar Galande, Pravara Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: abcd 2
Record Dates: First submitted 2010-09-17; First posted 2010-09-20 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2010-09

CONDITIONS: Primigravida in Labour Pains
Keywords: Analgesia, labour;; Analgesic techniques, epidural;; Drug delivery, intermittent bolus;; Anesthetics local, Bupivacaine;; Analgesics opioid, Fentanyl;
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bupivacaine-Fentanyl (3-15) (Active Comparator): Three millilitres of mixture of bupivacaine (0.125%) with fentanyl (2 µg/ml) injected through epidural catheter every 15 minutes as automated boluses.
  Interventions: Drug: Bupivacaine-Fentanyl Mixture
- Bupivacaine-Fentanyl (4-20) (Experimental): Four millilitres of mixture of bupivacaine (0.125%) with fentanyl (2 µg/ml) injected through epidural catheter every 20 minutes.
  Interventions: Drug: Bupivacaine-Fentanyl Mixture
- Bupivacaine-Fentanyl (6-30) (Experimental): Six millilitres of mixture of bupivacaine (0.125%) with fentanyl (2 µg/ml) injected through epidural catheter every 30 minutes.
  Interventions: Drug: Bupivacaine-Fentanyl Mixture

INTERVENTIONS:
Drug: Bupivacaine-Fentanyl Mixture — Three millilitres of mixture of bupivacaine (0.125%) with fentanyl (2 µg/ml) injected through epidural catheter every 15 minutes as automated boluses.
  Other Names: Bupivacaine-Fentanyl
  Arms: Bupivacaine-Fentanyl (3-15)
Drug: Bupivacaine-Fentanyl Mixture — Four millilitres of mixture of bupivacaine (0.125%) with fentanyl (2 µg/ml) injected through epidural catheter every 20 minutes.
  Other Names: Bupivacaine-Fentanyl
  Arms: Bupivacaine-Fentanyl (4-20)
Drug: Bupivacaine-Fentanyl Mixture — Six millilitres of mixture of bupivacaine (0.125%) with fentanyl (2 µg/ml) injected through epidural catheter every 30 minutes.
  Other Names: Bupivacaine-Fentanyl
  Arms: Bupivacaine-Fentanyl (6-30)

SUMMARY:
The purpose of this study is to determine how manipulation of the programmed intermittent time interval and volume influences total drug use, quality of analgesia, and patient satisfaction during maintenance of labor analgesia.

DETAILED DESCRIPTION:
Research for the ideal technique of maintaining epidural analgesia after the initial-level block is ongoing. Continuous infusion techniques, use of more dilute solutions , PCEA , and different techniques of PCEA like background dosing, none, fixed infusion as background, variable infusion (computer-integrated), programmed intermittent boluses (PIEBs) and automated mandatory boluses, have been used. Automated systems designed to administer a small bolus dose of anaesthetic at programmable intervals may combine the advantages of both manual bolus and continuous epidural infusion (CEI) systems.

Wong et al compared a PIEB (6 ml of bolus every 30 minutes) with CEI with the assumption that small frequent boluses may avoid wide fluctuations in sensory levels, commonly seen with traditional manually administered intermittent boluses and at the same time reduce the total anesthetic dose as in CEI. Chua and Sia showed that Pain scores were lower and the time to first manual epidural rescue bolus was longer in parturients assigned to intermittent boluses compared to continuous epidural infusion of the same solution in the intermittent group. Fettes and colleagues found that patients required a lower total drug dose and fewer manual bolus injections when epidural labor analgesia was maintained with automated intermittent boluses of ropivacaine compared to a continuous infusion. Solutions injected into the epidural space tend to spread more evenly when injected as a bolus, as compared to a continuous infusion. Furthermore, studies of epidural opioid analgesia suggest that epidural bolus administration of lipid soluble opioids (e.g., fentanyl) results in segmental spinal opioid analgesia, whereas continuous opioid epidural infusion results in systemic opioid analgesia. The analgesic effects of both epidural fentanyl infusion and epidural fentanyl bolus were evaluated using a volunteer, double blind, cross-over designs study. Taken together, the results of these studies suggest that further studies of automated intermittent bolus injections are indicated, in particular, studies of the optimal bolus time interval and volume. At one end of the spectrum, a short interval/low volume protocol may mimic a continuous infusion. At the other end of the spectrum, a long interval/large volume may negate the inherent safety of a continuous infusion. The purpose of the proposed study is to determine how manipulation of the programmed intermittent time interval and volume influences total drug use, quality of analgesia, and patient satisfaction during maintenance of labor analgesia.

Current pump technology does not support programmed intermittent bolus administration. The investigators encouraged the manufacturer to develop these features indigenously and incorporate them in presently available infusion pumps.

Methods:

Study will be carried out in randomly selected sixty uncomplicated full term pregnant patients, in active labour.

After written, informed, valid consent, and administration of five hundred millilitres of Ringer's lactate intravenously as a preload, epidural catheter will be inserted under aseptic conditions in an L2-L3 or L3-L4 space through 16 G Tuohy's needle. Epidural space will be identified through the loss-of-resistance technique. The catheter will be placed, cephaled, two spaces (3 to 4 cm) above the point of insertion.

Its position will be confirmed by administering a test dose of 3 ml of lignocaine (2%) with adrenaline.

A loading-dose mixture of 10 ml of bupivacaine (0.125%) and fentanyl (2 µg/ml) will be administered epidurally targeting initial sensory block to T 10 level .Additional doses of Inj.bupivacaine will be administered if required.

Infusion pump will be attached to the catheter and all patients will be randomly divided in three groups.

1. Group 3-15 : Three millilitres of mixture of bupivacaine (0.125%) with fentanyl (2 µg/ml) injected through epidural catheter every 15 minutes as automated boluses
2. Group 4-20: Four millilitres of mixture of bupivacaine (0.125%) with fentanyl (2 µg/ml) injected through epidural catheter every 20 minutes.
3. Group 6-30: Six millilitres of mixture of bupivacaine (0.125%) with fentanyl (2 µg/ml) injected through epidural catheter every 30 minutes.

Randomization will be carried out based on blocking. Blocks of size 3 with treatment allocation of 1:1:1 for group I, group II and group III will be created. A block of 3 patients will be assigned to one of the blocks created.

For blinding of patient as well observer, the settings of infusion pump will be hidden by covering it with cloth.

The level of sensory blockade will be tested by a pinprick method in midline and motor blockade will be tested with the modified Bromage scale used by Breen et al.

A single dose will be omitted if the sensory block goes higher than T7 or the motor blockade goes below score 4 as per the Bromage scale. Similarly additional top-ups of 3 ml of 0.125 % bupivacaine with fentanyl 2 micrograms / ml will be administered if patients get severe break through pain (VAS pain score > 3)

. Maternal parameters like pulse rate, blood pressure and respiratory rate will be monitored frequently. FHR will be monitored through tococardiography. Bearing-down ability will be assessed by asking the patients about the perception of the urge to bear down. Neonates will be assessed by Apgar score at 1 minute and 5 minutes after birth. The patients will be observed for any side effects or complications, such as pruritus, nausea and vomiting, hypotension, a headache, sedation and respiratory depression. Labour analgesic drug administration will be stopped after delivery and the duration of labour analgesia will be recorded. The total dose of bupivacaine and fentanyl will be calculated. The quality of analgesia will be assessed hourly. The patients will be asked about pain relief during the last hour and will be given scores as follows:

* 0 = No pain, pressure or tightening sensation
* 1 = Awareness of pressure or tightening sensation but not painful
* 2 = Slight pain or pressure sensation but not distressing
* 3 = Distressing pain or pressure sensation Even when the patients scored higher for a very short period, the higher score will be recorded for that hour. All the patients will be interviewed within 24 hours of delivery by an anaesthetist colleague who will unaware of the technique used and recorded a linear visual analogue scale (VAS) pain score on the patient's opinion about overall efficacy of analgesia. On this scale, 0 cm will indicate no pain and 10 cm will indicate worst pain. They will also ask about the level of their satisfaction regarding the quality of analgesia, which will be graded as 'excellent', 'good' and 'bad'.

Statistical analysis will be carried out with Stata 11.

ELIGIBILITY:
Inclusion Criteria:

* Full term women in spontaneous labor.
* Gestation greater than or equal to 37 weeks.
* Primigravida.
* Age group between 18 Years to 45 Years.
* ASA grade I or II
* Not having any complicated pregnancy
* Not having any systemic disorders.

Exclusion Criteria:

* Not willing for Epidural analgesia.
* Unwilling to get enrolled in this study.
* Systemic disorder like diabetes mellitus, hypertension and heart disease, spine deformity, blood coagulation disorder, bad obstetric history and foetal abnormity.
* Multiple-pregnancy or abnormal presentation.
* Complicated pregnancy like pregnancy induced hypertension, placenta previa, abruptio placenta.
* Cervical dilatation less than 2 or greater than 5 at time of initiation of neuraxial analgesia.
* Chronic analgesic medications
* Systemic opioid labor analgesia prior to the initiation of neuraxial labor analgesia.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Total epidural bupivacaine dose | 48 hours
  Labour analgesic drug administration will be stopped after delivery and the total dose of bupivacaine will be calculated.

SECONDARY OUTCOMES:
Demographics | 10 Minutes
  Age, Height,Weight
Quality of analgesia (Cumulative analgesia scores ) | Every Hour
  The quality of analgesia will be assessed hourly. The patients will be asked about pain relief during the last hour and will be given scores as follows:
  0 = No pain, pressure or tightening sensation
  1. = Awareness of pressure or tightening sensation but not painful
  2. = Slight pain or pressure sensation but not distressing
  3. = Distressing pain or pressure sensation Even when the patients scored higher for a very short period, the higher score will be recorded for that hour. Cumulative analgesia scores will be measured.
Level of analgesia (VAS score) | 48 hours
  All patients will be interviewed within 24 hours of delivery by an anaesthetist colleague who will unaware of the technique used and recorded a linear visual analogue scale (VAS) pain score on the patient's opinion about overall efficacy of analgesia. On this scale, 0 cm will indicate no pain and 10 cm will indicate worst pain.
Maternal satisfaction | 48 hours
  All the patients will be interviewed within 24 hours of delivery by an anaesthetist colleague who will unaware of the technique used and They will also ask about the level of their satisfaction regarding the quality of analgesia, which will be graded as 'excellent', 'good' and 'bad'.
No.of doses omitted | 48 hours
  A single dose will be omitted if the sensory block goes higher than T7 or the motor blockade goes below score 4 as per the Bromage scale.
No.of Additional top-ups required | 48 hours
  Additional top-ups of 3 ml of 0.125 % bupivacaine with fentanyl 2 micrograms / ml will be administered if patients get severe break through pain (VAS pain score > 3)
Duration of labour | 48 hours
  Labour analgesic drug administration will be stopped after delivery and the duration of labour will be recorded.
Maternal Safety | 48 hours
  Maternal parameters like pulse rate, blood pressure and respiratory rate will be monitored frequently.The patients will be observed for any side effects or complications, such as pruritus, nausea and vomiting, hypotension, a headache, sedation and respiratory depression.
Foetal Safety | 48 hours
  FHR will be monitored through tococardiography.Neonates will be assessed by Apgar score at 1 minute and 5 minutes after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Mandar V Galande, MBBS, Principal Investigator — Pravara Rural Hospital; Dr.Ramchandra V Shidhaye, MD DA, Principal Investigator — Pravara Rural Hospital; Dr.Devdas S Divekar, MD DA, Principal Investigator — Pravara Rural Hospital, Loni